CLINICAL TRIAL: NCT05990179
Title: Genomic Uniformed-Screening Against Rare Disease In All Newborns
Acronym: GUARDIAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Illumina, Inc. (Industry); GeneDx (Unknown); New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Rudolph L. Leibel, Professor of Pediatrics and Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AAAS9161
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Early Onset Genetic Conditions With Near Complete Penetrance
Keywords: Newborn screening; Genome sequencing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled in the study (Experimental): All newborns enrolled in the study will be evaluated.
  Interventions: Other: Genome sequencing-based newborn screening

INTERVENTIONS:
Other: Genome sequencing-based newborn screening — Dried blood spots collected at birth for routine newborn screening will be used for genome sequencing based screening of a defined set of conditions.

SUMMARY:
The goal of this study is to learn how genomic sequencing technology can be used to effectively expand the conditions screened on newborn screening. Newborn screening ensures equity and allows all babies to have the same chance at the healthiest life. Families will be invited to have their newborn baby screened for additional conditions beyond what all babies are screened for as part of the newborn screening public health program. Families can choose to be part of the study or choose not to be part of the study and just have the routine newborn screening test. Families will also be able to choose to learn about their baby's risk for conditions that have effective treatments available but are not on the routine newborn screening panel or also learn about conditions for which there is not currently FDA approved medications but for which medications are under development or for which early intervention services or treatment of seizures may improve the child's outcome. Families will be invited to the study shortly after the baby is born and will learn the decision not to participate, and we will interview a subset of parents who agree to be interviewed. Newborns who screen positive will be referred to appropriate providers for care and will be followed through review of electronic medical records and parental follow up via phone, text, postal mail or email.

DETAILED DESCRIPTION:
Newborn screening (NBS) is the process of screening all newborns for select conditions shortly after birth. This process reduces morbidity and mortality by the detection of medically actionable conditions in pre-symptomatic newborns. Approximately 1 in every 180 newborns is diagnosed with a condition through NBS. NBS is a public health service; every infant regardless of health insurance or ability to pay is tested. NBS ensures equity and allows all babies to have the same chance at the healthiest life. Effective NBS requires coordination and collaboration from multiple stakeholders - the parents, the hospital of birth, state department of health lab, the pediatrician, and the specialty referral center.

Conditions included on the NBS must fulfill several criteria: 1) significant clinical benefit for the newborn early in life including treatment administered within the first few years of life, 2) readiness of public health departments to effectively screen for the condition, and 3) feasibility of successful implementation of population screening. In the United States, screening of newborns is under the purview of state public health departments. Each state decides which disorders to screen, and expansions to each state's panel of screened conditions. The federal government also plays a role through the Secretary of Health and Human Services (HHS) Advisory Committee on Heritable Disorders in Newborns and Children (ACHDNC). With rapid improvements in screening technology, diagnostic testing, and treatments, conditions not previously screened through NBS are being considered. Expanding NBS through genome-wide sequencing (GS) will be the most flexible and cost-effective way to add to what is currently in use.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted to the well-baby nurseries from the recruiting hospitals
* Newborns born after 33 weeks of gestation
* Newborns whose parents are English, Mandarin, or Spanish speaking

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100000 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Enrollment Rate (percentage) | From study launch to end of enrollment (up to 5 years)
  Enrollment rate will be defined as: number of enrolled newborns / number of newborns approached by the research assistant.
Successful Sequencing Rate (percentage) | Up to 6 months after the end of enrollment
  Successful sequencing rate will be defined as: number of successful sequencing / number of enrolled newborns.
Screen Positive Rate (percentage) | Up to 6 months after the end of enrollment
  Screen positive rate will be defined as: number of newborns with a positive screening / number of successful sequencing.
True Positive Rate (percentage) | Up to 6 months after the end of enrollment
  True positive rate will be defined as: number of confirmed diagnosis / number of screen positive.

SECONDARY OUTCOMES:
Score on Decision Regret Scale | Up to 6 months after the end of enrollment
  The Decision Regret Scale measures distress or remorse after a health care decision. This 5-items scale ranges from 0 (no regrets - best outcome) to 100 (highest regret - worst outcome). Scores above 1 and below 25 are considered as an indication of mild regret. Scores above 25 are considered as an indication of moderate to severe regret.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy K. Chung, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Ziegler A, Koval-Burt C, Kay DM, Suchy SF, Begtrup A, Langley KG, Hernan R, Amendola LM, Boyd BM, Bradley J, Brandt T, Cohen LL, Coffey AJ, Devaney JM, Dygulska B, Friedman B, Fuleihan RL, Gyimah A, Hahn S, Hofherr S, Hruska KS, Hu Z, Jeanne M, Jin G, Johnson DA, Kavus H, Leibel RL, Lobritto SJ, McGee S, Milner JD, McWalter K, Monaghan KG, Orange JS, Pimentel Soler N, Quevedo Y, Ratner S, Retterer K, Shah A, Shapiro N, Sicko RJ, Silver ES, Strom S, Torene RI, Williams O, Ustach VD, Wynn J, Taft RJ, Kruszka P, Caggana M, Chung WK. Expanded Newborn Screening Using Genome Sequencing for Early Actionable Conditions. JAMA. 2025 Jan 21;333(3):232-240. doi: 10.1001/jama.2024.19662. PMID 39446378
- See also: GUARDIAN Study Website — https://guardian-study.org/